CLINICAL TRIAL: NCT02972827
Title: Comparison of the Accuracy of Monitoring Devices in Prediction of Fluid Responsiveness in Severe Sepsis and Septic Shock
Brief Title: Monitoring Devices in Prediction of Fluid Responsiveness in Severe Sepsis and Septic Shock
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Santa Barbara Cottage Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 15-21
Record Dates: First submitted 2016-10-30; First posted 2016-11-23 (Estimated); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: Severe Sepsis; Septic Shock
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NICOM/FloTrac (Experimental): 500-1000ml Crystalloid fluid challenge (normal saline or plasmalyte) to be given for positive passive leg raise test by either device, and also will be given at baseline, regardless of baseline PLR response.
  Interventions: Device: NICOM/FloTrac; Other: Crystalloid Fluid Challenge

INTERVENTIONS:
Device: NICOM/FloTrac — Use of noninvasive cardiac output and minimally invasive cardiac output monitors
Other: Crystalloid Fluid Challenge — 500-1000ml Normal Saline or Plasmalyte intravenous fluid bolus will be given at baseline, and following a positive passive leg raise response as defined by a 10% or greater increase in any of: stroke volume index, cardiac index, or pulse pressure, as measured by the NICOM or FloTrac Monitors.

SUMMARY:
Comparison of noninvasive cardiac output monitor (NICOM, Cheetah Medical) with Edwards FloTrac minimally-invasive cardiac output monitor in predicting fluid responsiveness in sepsis and septic shock.

DETAILED DESCRIPTION:
Study will evaluate ability of passive leg raise test to predict fluid responsiveness in patients in septic shock, on vasopressors, using both the NICOM and FloTrac devices. An increase in CI, SVI, or Pulse Pressure of >10% in response to the passive leg raise will be considered a positive passive leg raise test, and the same indicators will be considered a significant response to a fluid challenge with either crystalloids or colloids.Each device will be evaluated independently, but simultaneously.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients with severe sepsis or septic shock, who have arterial catheter placed with FloTrac monitor, with or without a central venous catheter.

Exclusion Criteria:

* Declination of consent
* Known allergy to adhesive
* Pregnancy
* Contraindication to raising legs or head to 45 degrees for 3 minute intervals

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Number of participants who have agreement or disagreement between passive leg raise response and subsequent intravenous fluid challenge | 15 minutes
  Positive passive leg raise response is defined as a 10% or greater increase in any of: stroke volume index, cardiac index, or pulse pressure following passive leg raise of 45 degrees for 3 minutes.
  Positive response to fluid challenge is defined as a 10% or greater increase in any of the same parameters following a 500ml or 1000 ml fluid challenge given over 10-15 minutes, using the same instrument, (NICOM or FloTrac). A negative response would be < 10% increase in these parameters using the same instrument

SECONDARY OUTCOMES:
Decrease in vasopressor dose, in response to fluid therapy guided by passive leg raise response using NICOM or Flotrac devices | 48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Santa Barbara Cottage Hospital, Santa Barbara, California, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-12-29): https://cdn.clinicaltrials.gov/large-docs/27/NCT02972827/Prot_SAP_000.pdf
  • Informed Consent Form (2016-12-29): https://cdn.clinicaltrials.gov/large-docs/27/NCT02972827/ICF_001.pdf